CLINICAL TRIAL: NCT02357940
Title: Clinical Trial to Evaluate the Tolerance of a Nighttime Moisturizing Balm on Babies and Adults With Mild to Moderate Atopic Dermatitis
Brief Title: Tolerance Evaluation of a Nighttime Moisturizing Balm on Babies and Adults With Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-140908134135-SBCT
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-11

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Eczema; Skin Irritation
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adult Tolerance Assessment (Experimental): Apply thin layer of experimental product to the affected skin areas at least 2 times per day and massage gently into skin
  Interventions: Drug: Experimental Product
- Baby (infants, toddlers, young children) Tolerance Assessment (Experimental): Apply thin layer of experimental product to the affected skin areas at least 2 times per day and massage gently into skin
  Interventions: Drug: Experimental Product

INTERVENTIONS:
Drug: Experimental Product — 1% Colloidal Oatmeal Balm
  Other Names: Eczema Moisturizing Balm

SUMMARY:
The purpose of this 14-day, two phase clinical study is to test the tolerance of a new over-the-counter moisturizing balm on subjects with eczema.

DETAILED DESCRIPTION:
At least 60 subjects will be enrolled to ensure 40 (10 adults and 30 babies) completed subjects. The tolerability of this formulation will be monitored in a small group of ten adult subjects with mild to moderate eczema prior to testing in babies. In Group A, adults will be asked to give their informed consent and an evaluation of inclusion/exclusion criteria will be performed at the site. After screening, all subjects will be asked not to use any skin treatments until the next clinic visit. Subjects will use the investigational product as indicated at least twice per day on the face - cheeks only, arms, legs and torso for 14 days. For both adults and babies, only the baseline measurements are collected at 5-10 minutes after first application, but not at Day 1, Day 7 and Day 14 visits. Babies from 6 to 36 months of age with mild to moderate eczema, who meet the eligibility criteria, will follow a similar testing directions in Group B of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race or ethnicity, 6 months to 36 months of age and/or 18 years and above.
2. Adult subjects only - Male or non-pregnant, non-lactating female agree to the contraceptive requirements (including female partners use of a highly effective form of birth control for 3 months.
3. Diagnosed as having Eczema.
4. Willing to stop the use of any non- assigned moisturizers and/or creams for the entire duration of the study.
5. Willing to not introduce any new fragrances (e.g. cleansers, lotions, perfumes, etc.), or in the household environment (e.g. room fresheners, cleansing agents, laundry detergents, etc.) for the duration of the study.
6. Willing to avoid excessive (more than 30 minutes) sun exposure without the use of their regular brand of sunscreen and protective clothing.
7. Willing to not enter/use hot tub or whirlpool bath for the duration of the study.
8. Willing to avoid the beach during the course of the study, and willing to document any activities at or in a swimming pool in the daily diary.

Exclusion Criteria:

1. Use of a therapeutic (over the counter or prescription) body wash that contains an active ingredient for eczema.
2. Adults Females who are pregnant (self-reported) or breastfeeding.
3. Participation in any clinical study within 30 days of Visit 1.
4. Atopic Dermatitis requiring systemic, super-potent (Class I) or potent (Class II or III) topical corticosteroids.
5. Requires greater than 2.0 mg/day inhaled or intranasal corticosteroids.
6. Subjects who exhibit clinically active bacterial, fungal, or viral skin infections or those who are susceptible to cutaneous infections.
7. Subjects who are currently on phototherapy.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amisha Parikh-Das, Ph.D., Study Director — Johnson & Johnson Consumer Inc. (J&JCI); Daniel Hogan, M.D., Principal Investigator — Hill-top Research Inc.; Ethlynn Schorr, M.D., Principal Investigator — TKL Research, Inc.
Locations (2):
- United States (2):
  - Hill-top Research, Inc, St. Petersburg, Florida
  - TKL Research Inc., Fair Lawn, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults: Adults - 1% Colloidal Oatmeal Balm
- Babies: Babies - 1% Colloidal Oatmeal Balm
Period: Overall Study
Arm/Group | Adults | Babies
Started | 9 | 32
Completed | 9 | 30
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Investigator's judgement | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adults | Babies | Total
Number analyzed (Participants) | 9 | 32 | 41
Age, Continuous [Mean (Standard Deviation); unit: months] | 400.0 (137.5) | 22.8 (8.89) | 105.6 (169.8)
Gender [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 3 | 19 | 22
Region of Enrollment [Number; unit: participants]
  USA | 9 | 32 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage With Erythema on the Face at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with erythema on the face at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 33.3 | 71.9
  0.5 | 55.6 | 6.3
  1 (Mild) | 11.1 | 21.9
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

2. Primary Outcome: Percentage With Erythema on the Arms at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with erythema on the arms at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 65.6
  0.5 | 22.2 | 9.4
  1 (Mild) | 0.0 | 18.8
  1.5 | 0.0 | 6.3
  2 (Moderate) | 22.2 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

3. Primary Outcome: Percentage With Erythema on the Legs at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with erythema on the legs at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 33.3 | 62.5
  0.5 | 33.3 | 9.4
  1 (Mild) | 11.1 | 25.0
  1.5 | 11.1 | 0.0
  2 (Moderate) | 11.1 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

4. Primary Outcome: Percentage With Erythema on the Torso at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with erythema on the torso at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 84.4
  0.5 | 22.2 | 0.0
  1 (Mild) | 22.2 | 12.5
  1.5 | 0.0 | 3.1
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

5. Primary Outcome: Percentage With Erythema on the Face at Baseline After Investigational Product Application
Description: Percentage of adults and babies with erythema on the face at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 75.0
  0.5 | 33.3 | 6.3
  1 (Mild) | 11.1 | 18.8
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

6. Primary Outcome: Percentage With Erythema on the Arms at Baseline After Investigational Product Application
Description: Percentage of adults and babies with erythema on the arms at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 68.8
  0.5 | 22.2 | 12.5
  1 (Mild) | 0.0 | 15.6
  1.5 | 0.0 | 3.1
  2 (Moderate) | 22.2 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

7. Primary Outcome: Percentage With Erythema on the Legs at Baseline After Investigational Product Application
Description: Percentage of adults and babies with erythema on the legs at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 68.8
  0.5 | 22.2 | 9.4
  1 (Mild) | 11.1 | 18.8
  1.5 | 11.1 | 3.1
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

8. Primary Outcome: Percentage With Erythema on the Torso at Baseline After Investigational Product Application
Description: Percentage of adults and babies with erythema on the torso at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 90.6
  0.5 | 22.2 | 0.0
  1 (Mild) | 22.2 | 3.1
  1.5 | 0.0 | 3.1
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

9. Primary Outcome: Percentage With Erythema on the Face at Day 1
Description: Percentage of adults and babies with erythema on the face at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 87.5
  0.5 | 44.4 | 3.1
  1 (Mild) | 0.0 | 9.4
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

10. Primary Outcome: Percentage With Erythema on the Arms at Day 1
Description: Percentage of adults and babies with erythema on the arms at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 78.1
  0.5 | 22.2 | 3.1
  1 (Mild) | 11.1 | 18.8
  1.5 | 11.1 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

11. Primary Outcome: Percentage With Erythema on the Legs at Day 1
Description: Percentage of adults and babies with erythema on the legs at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 75.0
  0.5 | 22.2 | 15.6
  1 (Mild) | 22.2 | 9.4
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

12. Primary Outcome: Percentage With Erythema on the Torso at Day 1
Description: Percentage of adults and babies with erythema on the torso at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 75.0
  0.5 | 33.3 | 3.1
  1 (Mild) | 22.2 | 18.8
  1.5 | 0.0 | 3.1
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

13. Primary Outcome: Percentage With Erythema on the Face at Day 7
Description: Percentage of adults and babies with erythema on the face at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 22.2 | 77.4
  0.5 | 55.6 | 6.5
  1 (Mild) | 22.2 | 16.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

14. Primary Outcome: Percentage With Erythema on the Arms at Day 7
Description: Percentage of adults and babies with erythema on the arms at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 33.3 | 77.4
  0.5 | 33.3 | 3.2
  1 (Mild) | 22.2 | 19.4
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

15. Primary Outcome: Percentage With Erythema on the Legs at Day 7
Description: Percentage of adults and babies with erythema on the legs at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 33.3 | 83.9
  0.5 | 55.6 | 3.2
  1 (Mild) | 0.0 | 12.9
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

16. Primary Outcome: Percentage With Erythema on the Torso at Day 7
Description: Percentage of adults and babies with erythema on the torso at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 33.3 | 87.1
  0.5 | 44.4 | 3.2
  1 (Mild) | 22.2 | 9.7
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

17. Primary Outcome: Percentage With Erythema on the Face at Day 14
Description: Percentage of adults and babies with erythema on the face at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 44.4 | 76.7
  0.5 | 55.6 | 6.7
  1 (Mild) | 0.0 | 16.7
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

18. Primary Outcome: Percentage With Erythema on the Arms at Day 14
Description: Percentage of adults and babies with erythema on the arms at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 44.4 | 83.3
  0.5 | 44.4 | 6.7
  1 (Mild) | 11.1 | 10.0
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

19. Primary Outcome: Percentage With Erythema on the Legs at Day 14
Description: Percentage of adults and babies with erythema on the legs at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 55.6 | 80.0
  0.5 | 33.3 | 10.0
  1 (Mild) | 0.0 | 6.7
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 3.3
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

20. Primary Outcome: Percentage With Erythema on the Torso at Day 14
Description: Percentage of adults and babies with erythema on the torso at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 44.4 | 86.7
  0.5 | 33.3 | 3.3
  1 (Mild) | 11.1 | 10.0
  1.5 | 0 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

21. Primary Outcome: Percentage With Edema on the Face at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with edema on the face at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 90.6
  0.5 | 33.3 | 6.3
  1 (Mild) | 0.0 | 3.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

22. Primary Outcome: Percentage With Edema on the Arms at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with edema on the arms at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 81.3
  0.5 | 0.0 | 6.3
  1 (Mild) | 11.1 | 9.4
  1.5 | 11.1 | 3.1
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

23. Primary Outcome: Percentage With Edema on the Legs at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with edema on the legs at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 22.2 | 81.3
  0.5 | 44.4 | 3.1
  1 (Mild) | 11.1 | 6.3
  1.5 | 0.0 | 3.1
  2 (Moderate) | 22.2 | 6.3
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

24. Primary Outcome: Percentage With Edema on the Torso at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with edema on the torso at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 84.4
  0.5 | 22.2 | 6.3
  1 (Mild) | 22.2 | 3.1
  1.5 | 11.1 | 6.3
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

25. Primary Outcome: Percentage With Edema on the Face at Baseline After Investigational Product Application
Description: Percentage of adults and babies with edema on the face at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 77.8 | 87.5
  0.5 | 22.2 | 9.4
  1 (Mild) | 0.0 | 3.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

26. Primary Outcome: Percentage With Edema on the Arms at Baseline After Investigational Product Application
Description: Percentage of adults and babies with edema on the arms at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 87.5
  0.5 | 11.1 | 3.1
  1 (Mild) | 0.0 | 6.3
  1.5 | 0.0 | 3.1
  2 (Moderate) | 22.2 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

27. Primary Outcome: Percentage With Edema on the Legs at Baseline After Investigational Product Application
Description: Percentage of adults and babies with edema on the legs at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 84.4
  0.5 | 22.2 | 3.1
  1 (Mild) | 11.1 | 6.3
  1.5 | 11.1 | 3.1
  2 (Moderate) | 11.1 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

28. Primary Outcome: Percentage With Edema on the Torso at Baseline After Investigational Product Application
Description: Percentage of adults and babies with edema on the torso at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 87.5
  0.5 | 0.0 | 3.1
  1 (Mild) | 22.2 | 6.3
  1.5 | 11.1 | 3.1
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

29. Primary Outcome: Percentage With Edema on the Face at Day 1
Description: Percentage of adults and babies with edema on the face at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 88.9 | 96.9
  0.5 | 11.1 | 0.0
  1 (Mild) | 0.0 | 3.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

30. Primary Outcome: Percentage With Edema on the Arms at Day 1
Description: Percentage of adults and babies with edema on the arms at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 90.6
  0.5 | 11.1 | 6.3
  1 (Mild) | 22.2 | 3.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

31. Primary Outcome: Percentage With Edema on the Legs at Day 1
Description: Percentage of adults and babies with edema on the legs at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 33.3 | 90.6
  0.5 | 44.4 | 6.3
  1 (Mild) | 11.1 | 0.0
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

32. Primary Outcome: Percentage With Edema on the Torso at Day 1
Description: Percentage of adults and babies with edema on the torso at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 90.6
  0.5 | 0.0 | 6.3
  1 (Mild) | 22.2 | 3.1
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

33. Primary Outcome: Percentage With Edema on the Face at Day 7
Description: Percentage of adults and babies with edema on the face at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 55.6 | 93.5
  0.5 | 33.3 | 6.5
  1 (Mild) | 11.1 | 0.0
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

34. Primary Outcome: Percentage With Edema on the Arms at Day 7
Description: Percentage of adults and babies with edema on the arms at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 44.4 | 93.5
  0.5 | 22.2 | 6.5
  1 (Mild) | 22.2 | 0.0
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

35. Primary Outcome: Percentage With Edema on the Legs at Day 7
Description: Percentage of adults and babies with edema on the legs at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 33.3 | 87.1
  0.5 | 55.6 | 6.5
  1 (Mild) | 0.0 | 3.2
  1.5 | 0.0 | 3.2
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

36. Primary Outcome: Percentage With Edema on the Torso at Day 7
Description: Percentage of adults and babies with edema on the torso at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 66.7 | 93.5
  0.5 | 0.0 | 3.2
  1 (Mild) | 11.1 | 3.2
  1.5 | 22.2 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

37. Primary Outcome: Percentage With Edema on the Face at Day 14
Description: Percentage of adults and babies with edema on the face at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 77.8 | 93.3
  0.5 | 22.2 | 0.0
  1 (Mild) | 0.0 | 6.7
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

38. Primary Outcome: Percentage With Edema on the Arms at Day 14
Description: Percentage of adults and babies with edema on the arms at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 55.6 | 83.3
  0.5 | 22.2 | 3.3
  1 (Mild) | 22.2 | 10.0
  1.5 | 0.0 | 3.3
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

39. Primary Outcome: Percentage With Edema on the Legs at Day 14
Description: Percentage of adults and babies with edema on the legs at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 44.4 | 80.0
  0.5 | 44.4 | 6.7
  1 (Mild) | 0.0 | 13.3
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

40. Primary Outcome: Percentage With Edema on the Torso at Day 14
Description: Percentage of adults and babies with edema on the torso at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 33.3 | 83.3
  0.5 | 44.4 | 13.3
  1 (Mild) | 0.0 | 3.3
  1.5 | 11.1 | 0.0
  2 (Moderate) | 11.1 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

41. Primary Outcome: Percentage With Scaling on the Face at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with scaling on the face at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 81.3
  0.5 | 33.3 | 9.4
  1 (Mild) | 0.0 | 6.3
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

42. Primary Outcome: Percentage With Scaling on the Arms at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with scaling on the arms at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 11.1 | 56.3
  0.5 | 33.3 | 3.1
  1 (Mild) | 33.3 | 28.1
  1.5 | 0.0 | 3.1
  2 (Moderate) | 22.2 | 6.3
  2.5 | 0.0 | 0
  3 (Severe) | 0.0 | 3.1

43. Primary Outcome: Percentage With Scaling on the Legs at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with scaling on the legs at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 0.0 | 34.4
  0.5 | 22.2 | 6.3
  1 (Mild) | 44.4 | 31.3
  1.5 | 22.2 | 12.5
  2 (Moderate) | 0.0 | 12.5
  2.5 | 11.1 | 0
  3 (Severe) | 0.0 | 3.1

44. Primary Outcome: Percentage With Scaling on the Torso at Baseline Before Investigational Product Application
Description: Percentage of adults and babies with scaling on the torso at baseline before investigational product application
Time Frame: At baseline before investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 22.2 | 71.9
  0.5 | 66.7 | 6.3
  1 (Mild) | 11.1 | 12.5
  1.5 | 0.0 | 6.3
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

45. Primary Outcome: Percentage With Scaling on the Face at Baseline After Investigational Product Application
Description: Percentage of adults and babies with scaling on the face at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 77.8 | 90.6
  0.5 | 22.2 | 6.3
  1 (Mild) | 0.0 | 0.0
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

46. Primary Outcome: Percentage With Scaling on the Arms at Baseline After Investigational Product Application
Description: Percentage of adults and babies with scaling on the arms at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 33.3 | 71.9
  0.5 | 44.4 | 12.5
  1 (Mild) | 22.2 | 12.5
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

47. Primary Outcome: Percentage With Scaling on the Legs at Baseline After Investigational Product Application
Description: Percentage of adults and babies with scaling on the legs at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 22.2 | 56.3
  0.5 | 66.7 | 21.9
  1 (Mild) | 11.1 | 18.8
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 3.1

48. Primary Outcome: Percentage With Scaling on the Torso at Baseline After Investigational Product Application
Description: Percentage of adults and babies with scaling on the torso at baseline after investigational product application
Time Frame: At baseline after investigational product application
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 55.6 | 78.1
  0.5 | 44.4 | 15.6
  1 (Mild) | 0.0 | 6.3
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

49. Primary Outcome: Percentage With Scaling on the Face at Day 1
Description: Percentage of adults and babies with scaling on the face at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 66.7 | 84.4
  0.5 | 33.3 | 6.3
  1 (Mild) | 0.0 | 9.4
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

50. Primary Outcome: Percentage With Scaling on the Arms at Day 1
Description: Percentage of adults and babies with scaling on the arms at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 44.4 | 75.0
  0.5 | 33.3 | 9.4
  1 (Mild) | 11.1 | 9.4
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 6.3
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

51. Primary Outcome: Percentage With Scaling on the Legs at Day 1
Description: Percentage of adults and babies with scaling on the legs at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 11.1 | 53.1
  0.5 | 66.7 | 18.8
  1 (Mild) | 11.1 | 18.8
  1.5 | 11.1 | 3.1
  2 (Moderate) | 0.0 | 3.1
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 3.1

52. Primary Outcome: Percentage With Scaling on the Torso at Day 1
Description: Percentage of adults and babies with scaling on the torso at Day 1
Time Frame: At Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 32
Percentage of participants
  0 (None) | 33.3 | 81.3
  0.5 | 66.7 | 6.3
  1 (Mild) | 0.0 | 9.4
  1.5 | 0.0 | 3.1
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

53. Primary Outcome: Percentage With Scaling on the Face at Day 7
Description: Percentage of adults and babies with scaling on the face at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 55.6 | 80.6
  0.5 | 44.4 | 3.2
  1 (Mild) | 0.0 | 16.1
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

54. Primary Outcome: Percentage With Scaling on the Arms at Day 7
Description: Percentage of adults and babies with scaling on the arms at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 44.4 | 74.2
  0.5 | 55.6 | 12.9
  1 (Mild) | 0.0 | 9.7
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 3.2
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

55. Primary Outcome: Percentage With Scaling on the Legs at Day 7
Description: Percentage of adults and babies with scaling on the legs at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 0.0 | 64.5
  0.5 | 44.4 | 16.1
  1 (Mild) | 44.4 | 12.9
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 3.2
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 3.2

56. Primary Outcome: Percentage With Scaling on the Torso at Day 7
Description: Percentage of adults and babies with scaling on the torso at Day 7
Time Frame: At Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 31
Percentage of participants
  0 (None) | 44.4 | 80.6
  0.5 | 44.4 | 12.9
  1 (Mild) | 11.1 | 6.5
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

57. Primary Outcome: Percentage With Scaling on the Face at Day 14
Description: Percentage of adults and babies with scaling on the face at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 66.7 | 83.3
  0.5 | 33.3 | 6.7
  1 (Mild) | 0.0 | 10.0
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

58. Primary Outcome: Percentage With Scaling on the Arms at Day 14
Description: Percentage of adults and babies with scaling on the arms at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 33.3 | 80.0
  0.5 | 44.4 | 0.0
  1 (Mild) | 11.1 | 13.3
  1.5 | 0.0 | 0.0
  2 (Moderate) | 11.1 | 6.7
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

59. Primary Outcome: Percentage With Scaling on the Legs at Day 14
Description: Percentage of adults and babies with scaling on the legs at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 22.2 | 70.0
  0.5 | 44.4 | 6.7
  1 (Mild) | 22.2 | 20.0
  1.5 | 11.1 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 3.3

60. Primary Outcome: Percentage With Scaling on the Torso at Day 14
Description: Percentage of adults and babies with scaling on the torso at Day 14
Time Frame: At Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Adults | Babies
Number analyzed (Participants) | 9 | 30
Percentage of participants
  0 (None) | 33.3 | 80.0
  0.5 | 66.7 | 13.3
  1 (Mild) | 0.0 | 6.7
  1.5 | 0.0 | 0.0
  2 (Moderate) | 0.0 | 0.0
  2.5 | 0.0 | 0.0
  3 (Severe) | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Day 14 ± 2 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected at each study visit through Visit 5 (Day 14 ± 2 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | Adults | Babies
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/32
Other Adverse Events (participants affected / at risk) | 1/9 | 0/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adults (N=9) | Babies (N=32)
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators agreed not to publish the study results without prior sponsor approval.